CLINICAL TRIAL: NCT04052399
Title: Improving Insulin Sensitivity by Non-invasive Brain Stimulation- Feasibility Study
Brief Title: Improving Insulin Sensitivity by Non-invasive Brain Stimulation in Persons With Insulin Resistance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Collaborators: German Center for Diabetes Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 243/2019BO1
Record Dates: First submitted 2019-08-06; First posted 2019-08-09 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2019-08

CONDITIONS: Insulin Resistance; Transcranial Direct Current Stimulation
MeSH Terms: conditions — Insulin Resistance | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anodal tDCS (Active Comparator): Anodal tDCS of the lateral hypothalamus-cognitive or medial hypothalamus-cognitive network (2 conditions)
  Interventions: Device: anodal transcranial direct current stimulation
- Cathodal tDCS (Active Comparator): Cathodal tDCS of the lateral hypothalamus-cognitive or medial hypothalamus-cognitive network (2 conditions)
  Interventions: Device: cathodal transcranial direct current stimulation
- Sham stimulation (Placebo Comparator): Single blind sham stimulation (ramp-up ramp-down stimulation will be applied for 30 seconds in order to simulate the active condition without any further continuous administration of current)
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: anodal transcranial direct current stimulation — Anodal tDCS of the lateral hypothalamus-cognitive or medial hypothalamus-cognitive network.
  The total injected current will never go beyond 4 milliamp, which will be split among the different stimulation electrodes.
  Other Names: anodal tDCS
  Arms: Anodal tDCS
Device: cathodal transcranial direct current stimulation — Cathodal tDCS of the lateral hypothalamus-cognitive or medial hypothalamus-cognitive network.
  The total injected current will never go beyond 4 milliamp, which will be split among the different stimulation electrodes.
  Other Names: cathodal tDCS
  Arms: Cathodal tDCS
Device: transcranial direct current stimulation — Single blind sham stimulation (ramp-up ramp-down stimulation will be applied for 30 seconds)
  Other Names: tDCS
  Arms: Sham stimulation

SUMMARY:
Efforts in curing and preventing obesity and type 2 diabetes (T2D) have been elusive thus far. One reason for that is the lack of understanding of the role of the brain in the development and treatment of the disease. Insulin action in the brain is appreciated to play a vital role in the pathophysiology of T2D, influencing eating behavior, cognition and peripheral metabolism. Whether brain insulin resistance is a cause or consequence of prediabetes is not yet fully understood. Hence, in this project the investigators want to develop a novel tool to treat and prevent type 2 diabetes and to delineate brain mechanisms of insulin resistance in humans. For this purpose, transcranial direct current stimulation (tDCS) will be implemented, which is a powerful tool to stimulate brain networks. In recent studies, it was shown that the hypothalamus is part of a brain network including higher cognitive regions that is particularly vulnerable to insulin resistance. Furthermore, the central insulin response in this network predicted food craving and hunger. The investigators hypothesize that stimulating the hypothalamus-cognitive network will enhance insulin sensitivity and reduce food intake, food craving and hunger. Furthermore, the project will provide the unique opportunity to investigate novel mechanisms of insulin resistance in participants who have been extensively metabolically characterized.

DETAILED DESCRIPTION:
Objectives The overarching aim of the study is to stimulate the hypothalamus-cognitive brain network to improve insulin sensitivity and eating behavior.

Specific Objectives- Feasibility study:

1. Implement resting-state functional magnetic resonance imaging to identify individual medial and lateral hypothalamic cognitive functional networks.
2. Evaluate and test different non-invasive brain stimulation paradigms by tDCS to stimulate lateral and medial hypothalamus cognitive network on eating behavior and metabolism.

   20 participants with overweight and obesity will receive five different tDCS stimulation protocols on five separate days (separated by one week) in a single-blind cluster-randomized order to reduce sequence effects. Optimal stimulation sites are assessed of the lateral and medial hypothalamus-cognitive network based on a modelling approach. Since this is the first study to stimulate the hypothalamus-cognitive network, excitatory as well as inhibitory stimulation is used. To reduce the number of conditions, participant are randomized based on the three main conditions: sham stimulation, anodal and cathodal stimulation. Medial hypothalamus-cognitive network versus lateral hypothalamus-cognitive network stimulation are pseudo-randomised.

   Participants will come in the morning, after an overnight fast, to receive a 20 min non-invasive brain stimulation, using tDCS. During the stimulation, participants will perform a stop-signal task on an tablet.

   Subsequently, participants will receive a breakfast buffet. The caloric intake from fat, carbohydrates and protein will be documented. Subjective feeling of hunger and food craving will be assessed using a visual analogue scale before stimulation, directly after stimulation and after breakfast. Food pictures will be rated on a laptop for taste and healthiness.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 25.5 and 35 kg/m2
* Age between 20 to 60 years of age
* Criteria for prediabetes:

Fasting plasma glucose (PG) 100 mg/dL (5.6 mmol/L) to 125 mg/dL (6.9 mmol/L) (impaired fasting glucose) OR 2-h PG during 75-g oral glucose tolerance test 140 mg/dL (7.8 mmol/L) to 199 mg/dL (11.0 mmol/L) (impaired glucose tolerance) OR HbA1c 5.7-6.4% (39-47 mmol/mol)

Exclusion Criteria:

* Insufficient knowledge of the German language
* Persons who cannot legally give consent
* Pregnancy or lactation
* History of severe mental or somatic disorders including neurological diseases (incl. epileptic seizures)
* Taking psychotropic drugs
* Previous bariatric surgery
* Acute infection within the last 4 weeks
* Hemoglobin values less than 12g/dl for women, less than 14 g/dl for men
* Current participation in a lifestyle intervention study or a pharmaceutical study
* Contradictions to a MRI measurement (e.g. metal implants)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-11-04 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Caloric intake (kcal) | 1 hour after tDCS
  The investigators will assess free-choice, ad libitum food intake from a standardized breakfast buffet. The caloric intake from fat, carbohydrates and protein will be documented.
Change in subjective feeling of hunger and food craving | 5 minutes before tDCS, 10 min after tDCS and 10 min after breakfast
  On a visual analogue scale, subjective feeling of hunger and food craving will be assessed using a questionnaire.

SECONDARY OUTCOMES:
Response inhibition | 20 minutes during tDCS
  To measure the performance during the stop-signal task (i.e. response inhibition) direction errors, proportion of successful stops, reaction time on Go trials, and stop signal reaction time (SSRT) will be measured.
Tastiness and healthiness rating of food stimuli | 10 minutes task after breakfast
  Using a computer based task, participants rate food pictures of low caloric and high caloric foods and snacks on a 5-point scale based on subjective tastiness and healthiness (1=not at all tasty/very unhealthy, 2=not tasty/unhealthy, 5 very tasty/healthy).
Food choice | 10 minutes task after rating of food stimuli
  Using a computer based task, participants have to choose food items they preferred to eat compared to a reference food on a 5-point choice scale. The reference (or "neutral") food item is individually determined based the health and taste rating.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Kullmann, PhD, Principal Investigator — University Hospital Tübingen
Locations (1):
- University Clinic Tübingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No